CLINICAL TRIAL: NCT05237856
Title: The Use of End Tidal CO2 and Integrated Pulmonary Index to Predict Post Spinal Hypotension in Cesarean Section
Brief Title: The Use of Integrated Pulmonary Index During Cesarean Section Under Spinal Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Assistant professor, Selcuk University
Other Study IDs: IPI
Record Dates: First submitted 2022-01-07; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Intraoperative Hypotension
Keywords: cesarean, hypotension, ETCO2, integrated pulmonary index
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Capnometry Monitorization — After spinal anesthesia, a non-invasive nasal cannula will be applied to the patient, ETCO2 and IPI values will be continuously measured and recorded from this cannula with a capnometry device.

SUMMARY:
Postspinal hypotension (PSH) is a common side effect with an incidence of 15.3 to 33% that can result in organ hypoperfusion and ischemic events. In pregnant patients, this incidence may increase to 70% and severe PSH increases the risk of maternal and fetal complications. Therefore, it is extremely important for anesthesiologists to recognize PSH early and treat it quickly during cesarean sections.

Integrated pulmonary index (IPI) is an algorithm that has been used recently. IPI takes into account four parameters: respiratory rate, end tidal CO2, heart rate and O2 saturation. Capnography device measuring IPI can continuously monitor and display the patient's respiratory status in a single digit range from 1-10. This index value can be observed continuously on the monitor as digital data or as a waveform. "10" indicates a normal respiratory condition, while "1" indicates that the patient requires immediate intervention. The relationship between values and the patient status is evaluated as follows; 10 = Normal, 8-9 = Normal range, 7 = Near normal range; Requires attention, 5-6 = Requires attention and may require intervention, 3-4 = Requires intervention, 1-2 = Requires immediate intervention.

IPI monitorization is mostly used during sedation (gastroscopy, cardioversion), intensive care units (for adjusting mechanical ventilator settings, monitoring the weaning process).

As a result, IPI monitoring has attracted attention because it allows non-invasive, dynamic and real-time measurement, reflects respiratory status with high specificity and sensitivity, and enables respiratory problems to be detected earlier.

End tidal CO2, which is one of the 4 parameters that IPI value takes into account, is a parameter that can be used to evaluate the effectiveness of ventilation, but is also related to cardiac output (CO) because the delivery of CO2 to the pulmonary system depends on it. Studies have shown that ETCO2 value correlatively decreases when CO decrease, in cases such as hypotension and hypovolemia.

We think that ETCO2 will decrease due to pulmonary hypoperfusion in post spinal hypotension and it may cause a change in IPI value. In our study, we will monitor patients who are scheduled for cesarean section under spinal anesthesia with a capnometry device and we will try to determine the significance of IPI monitorization in predicting hypotension.

DETAILED DESCRIPTION:
Patients who underwent cesarean section under spinal anesthesia and who agreed to participate in the study will be included in the study.

Demographic data of the patients (age, gender, weight, concomitant diseases, etc.) will be recorded.

After spinal anesthesia, a non-invasive nasal cannula will be inserted into the patients, and ETCO2 and IPI values will be continuously measured and recorded from this cannula with a capnometry device.

As is routinely done, blood pressure will be measured at 2-minute intervals after spinal anesthesia is administered.

The non-invasive blood pressure value measured before spinal anesthesia will be taken as the baseline value, and a decrease of 20% or more in this value or a decrease in systolic blood pressure below 100 mmHg will be considered hypotension.

The correlation between the developing hypotension and the End tidal CO2 and IPI measurements will be examined.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II pregnants who will undergo cesarean section under spinal anesthesia

Exclusion Criteria:

* ASA III- IV Pregnants.
* Pregnants with chronic respiratory disorder.
* Pregnants who will undergo cesarean section under emergency conditions.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnants above the age of 18 who will undergo cesarean section under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
noninvasive blood pressure | 20 minutes
  hypotension:20% reduction in basal blood pressure measurement,
Integrated pulmoner index (IPI) | 20 minutes
  requires intervention: IPI value < 7,
end-tidal carbon dioxide (ETCO2) | 20 minutes
  hypoperfusion: ETCO2 value < 35 mmHg